CLINICAL TRIAL: NCT00308711
Title: A Multi-center, Randomized, Double-blind Phase III Study of the Efficacy and Safety of the Misoprostol Vaginal Insert Compared to Cervidil for Women Requiring Cervical Ripening and Induction of Labor (The MVP Study).
Brief Title: Safety/Efficacy Study Comparing the Misoprostol Vaginal Insert to Cervidil for Cervical Ripening and Induction of Labor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Miso-Obs-004
Record Dates: First submitted 2006-03-27; First posted 2006-03-30 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Ripening; Labor, Induced
Keywords: Cervical ripening; Induction of labor; Dinoprostone vaginal insert; Cervidil; Misoprostol vaginal insert; Modified Bishop's Score; PGE2; PGE1; Uterine Hyperstimulation; Cesarean section
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MVI 100 (Experimental): Misoprostol vaginal insert 100 mcg over 24h
  Interventions: Drug: Misoprostol vaginal insert 100 mcg
- MVI 50 (Experimental): Misoprostol vaginal insert 50 mcg over 24h
  Interventions: Drug: Misoprostol vaginal insert 50 mcg
- Cervidil 10 mg vaginal insert (Active Comparator): Cervidil 10 mg over 24h
  Interventions: Drug: Dinoprostone vaginal insert (Cervidil)

INTERVENTIONS:
Drug: Misoprostol vaginal insert 100 mcg — Hydrogel polymer intravaginal insert with retrieval system. One insert is to remain in the posterior fornix of the vagina until removed for one of the following conditions: onset of active labor; maternal/fetal complication, e.g. non-reassuring fetal heart rate. Record if the insert falls out prior to meeting one of the first two criteria. In no case is the insert to remain in place longer than 24h.
  Other Names: Misopess(TM)
  Arms: MVI 100
Drug: Misoprostol vaginal insert 50 mcg — Hydrogel polymer intravaginal insert with retrieval system. One insert is to remain in the posterior fornix of the vagina until removed for one of the following conditions: onset of active labor; maternal/fetal complication, e.g. non-reassuring fetal heart rate. Record if the insert falls out prior to meeting one of the first two criteria. In no case is the insert to remain in place longer than 24h.
  Other Names: Misopess(TM)
  Arms: MVI 50
Drug: Dinoprostone vaginal insert (Cervidil) — Hydrogel polymer intravaginal insert with retrieval system. One insert is to remain in the posterior fornix of the vagina until removed for one of the following conditions: onset of active labor; maternal/fetal complication, e.g. non-reassuring fetal heart rate. Record if the insert falls out prior to meeting one of the first two criteria. In no case is the insert to remain in place longer than 24h.
  Other Names: Propess(R); 10 mg dinoprostone vaginal insert
  Arms: Cervidil 10 mg vaginal insert

SUMMARY:
The purpose of this study is to determine whether the misoprostol vaginal insert (50 mcg and 100 mcg) can safely and effectively speed time to vaginal delivery compared to Cervidil (R) in women who need to have cervical ripneing and induction of labor.

DETAILED DESCRIPTION:
Induction of labor is required in approximately 20% of pregnant women. Although contractions can be brought on by oxytocin ("pitocin"), some women need help in softening the cervix, or mouth of the womb (uterus), before oxytocin can be started. Prostaglandins have been shown to ripen, or soften, the cervix; at present, the only prostaglandin approved for marketing by FDA for this purpose is dinoprostone. Dinoprostone can be delivered in several ways; one method is to use a polymer vaginal insert that slowly releases the dinoprostone directly to the cervical tissues. This product is called Cervidil (R) and has been marketed for more than 10 years in the United States. Misoprostol is another form of prostaglandin that is approved for protecting the stomach and intestinal lining for patients taking NSAIDs. Misoprostol has also been used by many obstetricians for cervical ripening and inducing contractions, but, it is not approved by FDA for this purpose.

The same company that makes the Cervidil polymer insert has made an insert that will slowly release misoprostol. This study will determine whether this investigational insert containing misoprostol will decrease time to vaginal delivery compared to Cervidil. Two different doses of misoprostol will be tested (50 micrograms and 100 micrograms); each vaginal insert will gradually release a small, controlled amount of misoprostol over up to 24 hours.

Comparator: The Cervidil (R) vaginal insert containing dinoprostone will be the comparator in this study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 36 weeks gestation requiring cervical ripening and induction of labor

Exclusion Criteria:

* No uterine scar (no previous delivery by cesarean section)
* No multiple gestation
* No condition that disallows use of prostaglandins for induction of labor
* No more than 3 previous vaginal births beyond 24 weeks gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1308 (Actual)
Dates: Start 2006-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director
Locations (52):
- United States (49):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Maricopa Medical Center, Phoenix, Arizona
  - Arizona Wellness Center for Women, Phoenix, Arizona
  - Tuscon Medical Center, Tucson, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - UCI Medical Center, Orange, California
  - Santa Clara Valley Medical Center, San Jose, California
  - Christiana Care Health System, Newark, Delaware
  - Bayfront Medical Center, St. Petersburg, Florida
  - University of Florida Health Sciences Center, Tampa, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Northside Hospital, Alpharetta, Georgia
  - Hurley Medical Center, Flint, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - St. Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Morristown Memorial Hospital, Morristown, New Jersey
  - University of New Mexico Medical Center, Albuquerque, New Mexico
  - United Health Services Hospitals, Inc., Johnson City, New York
  - Winthrop-South Nassau University Health Center, Mineola, New York
  - NYU School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Women's Health Alliance, Winston-Salem, North Carolina
  - University of Cincinnati Holmes Hospital, Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Center for Maternal-Fetal Medicine, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Medical Center, Allentown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Greenville Hospital System, Greenville, South Carolina
  - Trident Health System, North Charleston, South Carolina
  - Erlanger Hospital, Chattanooga, Tennessee
  - University of Tennesse Medical Center, Knoxville, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Methodist Charlton Medical Center, Dallas, Texas
  - University of Texas Health Sciences Center at Houston, Houston, Texas
  - Kings Daughters Clinic, Temple, Texas
  - McKay-Dee Hospital, Ogden, Utah
  - St. Mark's Hospital, Salt Lake City, Utah
  - University of Utah Health Science Center, Salt Lake City, Utah
  - Jordan Valley Hospital, West Jordan, Utah
  - Pioneer Valley Hospital, West Valley City, Utah
  - Overlake Hospital Medical Center, Bellevue, Washington
  - Saint Clare's Hospital, Weston, Wisconsin
- Canada (3):
  - Women's Health Centre/General Hospital/Eastern Health, St. John's, Newfoundland and Labrador
  - IWK Health Centre and Dalhousie University, Halifax, Nova Scotia
  - University of Saskatchewan Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Castaneda CS, Izquierdo Puente JC, Leon Ochoa RA, Plasse TF, Powers BL, Rayburn WF. Misoprostol dose selection in a controlled-release vaginal insert for induction of labor in nulliparous women. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 2):1071-5. doi: 10.1016/j.ajog.2005.06.072. PMID 16157114
- [Background] Rayburn WF, Powers BL, Plasse TF, Carr D, Di Spirito M. Pharmacokinetics of a controlled-release misoprostol vaginal insert at term. J Soc Gynecol Investig. 2006 Feb;13(2):112-7. doi: 10.1016/j.jsgi.2005.10.004. PMID 16443504
- [Background] Ewert K, Powers B, Robertson S, Alfirevic Z. Controlled-release misoprostol vaginal insert in parous women for labor induction: a randomized controlled trial. Obstet Gynecol. 2006 Nov;108(5):1130-7. doi: 10.1097/01.AOG.0000239100.16166.5a. PMID 17077234
- [Result] Wing DA; Misoprostol Vaginal Insert Consortium. Misoprostol vaginal insert compared with dinoprostone vaginal insert: a randomized controlled trial. Obstet Gynecol. 2008 Oct;112(4):801-12. doi: 10.1097/AOG.0b013e318187042e. PMID 18827122
- [Result] Pevzner L, Rayburn WF, Rumney P, Wing DA. Factors predicting successful labor induction with dinoprostone and misoprostol vaginal inserts. Obstet Gynecol. 2009 Aug;114(2 Pt 1):261-267. doi: 10.1097/AOG.0b013e3181ad9377. PMID 19622986
- [Derived] Hawkins JS, Stephenson M, Powers B, Wing DA. Diabetes mellitus: an independent predictor of duration of prostaglandin labor induction. J Perinatol. 2017 May;37(5):488-491. doi: 10.1038/jp.2016.270. Epub 2017 Jan 26. PMID 28125096
- [Derived] Brennan MC, Pevzner L, Wing DA, Powers BL, Rayburn WF. Retention of dinoprostone vaginal insert beyond 12 hours for induction of labor. Am J Perinatol. 2011 Jun;28(6):479-84. doi: 10.1055/s-0030-1271208. Epub 2011 Jan 11. PMID 21225563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject entered 26 April 2006; last subject completed 07 August 2007; 49 hospitals entered subjects requiring cervical ripening prior to induction of labor.
Groups:
- Misoprostol Vaginal Insert (MVI) 100: Misoprostol vaginal insert 100 mcg over a period of up to 24 h
- Misoprostol Vaginal Insert (MVI) 50: Misoprostol vaginal insert 50 mcg over a period of up to 24 h
- Cervidil 10 mg Vaginal Insert: Cervidil 10 mg vaginal insert over a period of up to 24h
Period: Overall Study
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Started | 428 | 444 | 436
Completed | 426 | 440 | 431
Not Completed | 2 | 4 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Baby not born within 7 days of treatment | 1 | 2 | 2
Not completed — Subject incarcerated, data not allowed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert | Total
Number analyzed (Participants) | 428 | 444 | 436 | 1308
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 428 | 444 | 436 | 1308
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.2 (5.9) | 26.9 (6.2) | 26.0 (5.7) | 26.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 428 | 444 | 436 | 1308
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 413 | 427 | 419 | 1259
  Canada | 15 | 17 | 17 | 49
Parity [Number; unit: participants] — Nulliparaous = no previous vaginal delivery prior to 24 wks gestation Parous = at least one previous vaginal delivery after 24 weeks
  participants
    Nulliparous | 267 | 275 | 270 | 812
    Parous | 161 | 169 | 166 | 496
modified Bishop score (mBS) [Mean (Standard Deviation); unit: Units on a scale of 0 (low) to 12 (most)] — The mBS measures cervical softness. There are five elements assessed during a vaginal examination. Maximum mBS is 12: 0 to 3 for Dilation, 0 to 3 for Station, 0 to 2 for Consistency, 0 to 1 for Position, and 0 to 3 for Length of Cervix. A score of zero is a long, closed, thick firm cervix; a score of 12 indicates thin, completely soft, 100% effaced cervix.
  Units on a scale of 0 (low) to 12 (most) | 2.69 (1.1) | 2.74 (1.1) | 2.73 (1.1) | 2.72 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Minutes From Drug Insertion to Vaginal Delivery
Description: Interval between time/date of insertion of study drug and time/date of neonate birth. This is a time-to-event analysis, there is no set time for the assessment. The endpoint occurs when the baby is born. 48 hours can be used as an approximate interval by which time most of the babies have been delivered.
Time Frame: 2880 minutes
Population: This analysis is for time to vaginal delivery (interval from insertion of study drug into the vagina to the delivery of the neonate); patients delivered by cesarean section were censored from this time-to-event analysis using the longest interval for all participants from insertion of study drug to cesarean section delivery of neonate.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
minutes | 1595.5 [1469 to 1739] | 2127 [1977 to 2253] | 1649.5 [1509 to 1824]
Statistical Analysis 1: Comparison: Misoprostol Vaginal Insert (MVI) 100 vs Cervidil 10 mg Vaginal Insert; Null hypothesis was that there would be no difference in time to vaginal delivery for MVI 100 compared to time to vaginal delivery for Cervidil; Test type: Superiority or Other; p = 0.974, Log Rank — The a priori threshold for statistical significance was 0.05; Kaplan-Meier = 1595.5 — This was a Kaplan-Meier analysis of median time to vaginal delivery. Cervidil was compared separately to MVI 100 and MVI 50
Statistical Analysis 2: Comparison: Misoprostol Vaginal Insert (MVI) 50 vs Cervidil 10 mg Vaginal Insert; Test type: Superiority or Other; p = 0.011, Log Rank; Cox Proportional Hazard = 1977, 95% CI [1977 to 2253]

2. Primary Outcome: Percentage of Participants With a Cesarean Section Delivery
Description: Percentage of participants with cesarean delivery after study drug was administered. There is no set assessment time or date as the woman's labor may last hours or days.
Time Frame: 2880 minutes
Measure: Number; unit: Percentage of participants
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
Percentage of participants | 28 [23.6 to 32.3] | 28 [23.9 to 32.4] | 26 [22.3 to 30.8]
Statistical Analysis 1: Comparison: Misoprostol Vaginal Insert (MVI) 100 vs Cervidil 10 mg Vaginal Insert; Test type: Non-Inferiority or Equivalence — Non-inferiority (NI) margin was within 15% relative to the rate of cesarean section for the comparator (Cervidil 10 mg dinoprostone vaginal insert); p = 0.64, Fisher Exact; Cox Proportional Hazard = 27.8, 95% CI [23.61 to 32.31]
Statistical Analysis 2: Comparison: Misoprostol Vaginal Insert (MVI) 50 vs Cervidil 10 mg Vaginal Insert; Test type: Non-Inferiority or Equivalence — Non-inferiority margin was rate of cearean section within 15% of Cervidil rate; p = 0.59, Fisher Exact; Cox Proportional Hazard = 28.0, 95% CI [23.86 to 32.42]

3. Secondary Outcome: Percentage of Participants With Maternal/Fetal, Maternal (Post-Partum), and Neonatal Adverse Events
Description: This outcome reports the percentage of adverse events in each treatment arm spontaneously reported or observed during the study. The intrapartum period (mother is still pregnant) is called the "Maternal/Fetal" period; once the baby has been born, adverse events are assessed separately for the mother (Post Partum) and the baby (Neonatal). The number of adverse events was assessed separately for each of the three periods.
Time Frame: 96 hours
Population: Analysis was based on intention to treat, i.e., all subjects who had the insert placed in the vagina.
Measure: Number; unit: Percentage of participants
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
Percentage of participants
  Maternal/Fetal | 65 | 64 | 65
  Maternal (Post-Partum) | 29 | 26 | 27
  Neonatal | 29 | 24 | 27

4. Secondary Outcome: Percentage of Participants With Pre-Delivery Oxytocin Use
Description: Incidence in each treatment group of need for oxytocin for pre-delivery induction or augmentation of labor.
Time Frame: 2880 minutes
Population: This analysis included all participants exposed to study drug and for whom there was data available regarding whether oxytocin was used pre-delivery.
Measure: Number; unit: Percentage of participants
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
Percentage of participants | 68.5 | 80.8 | 69.0

5. Secondary Outcome: Percentage of Participants With Cervical Ripening Success Based On Modified Bishop Score (mBS) 12 Hours After Administration of Vaginal Insert
Description: Measured the percentage of participants who achieved success on the mBS. This composite score is based on the mBS and vaginal delivery and it is measured 12 hours after insertion of the study drug. The mBS has a score of 0 when the cervix is not ripe and a score of 12 when completely ripened. The 12 hour score is compared to baseline. Using the mBS, assess at 12 hours whether each subject has met any of the following three criteria: 1) has improved (increased) the mBS by at least 3 points from baseline; 2) has reached a score of at least 6 on the mBS; or 3) has acheived a vaginal delivery.
Time Frame: 12 hours
Measure: Number; unit: Percentage of Participants
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
Percentage of Participants | 59 (3.15) | 50 (2.8) | 60 (3.3)

6. Secondary Outcome: Minutes to Onset of Active Labor
Description: Interval from insertion of study drug to onset of active labor, defined as at least three contractions in a ten-minute period of at least moderate intensity and resulting in cervical change such as dilatation or effacement; OR at least 4 cm cervical dilatation achieved after progressive change in dilatation.
Time Frame: 2880 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
minutes | 1032.5 (627.2) | 1343.7 (692.0) | 1005.2 (667.1)

7. Secondary Outcome: Minutes to Rupture of Membranes (ROM)
Description: Interval from study drug insertion to ROM.
Time Frame: 2880 minutes
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
minutes | 1285.0 [906.0 to 2208.0] | 1364.0 [1048 to 2491] | 1123 [915 to 1580]

8. Secondary Outcome: Duration of Stay in Minutes in Labor and Delivery Suite
Description: Minutes in Labor and Delivery (L & D) suite starting from insertion of the study drug to discharge from L & D to post partum care.
Time Frame: 5760 minuts
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
minutes | 1683.6 (811) | 2010 (850) | 1729 (862)

9. Secondary Outcome: Days in Hospital for Mother and Neonate
Description: Duration of stay in hospital for mother and neonate starting with insertion of the study drug and ending with discharge from the hospital.
Time Frame: 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Number analyzed (Participants) | 426 | 440 | 431
days
  Mother | 4.5 (1.24) | 4.7 (1.1) | 4.5 (1.3)
  Neonate | 3.6 (1.8) | 3.5 (1.2) | 3.6 (1.6)

ADVERSE EVENTS:
Time Frame: 96 hours
Description: Adverse event data were collected during the hospital period only. One subject in the MVI 50 group was incarcerated; her information was not permitted to be used for data analysis, therefore all results are based on 443 subjects for this treatment groups.
Arm/Group | Misoprostol Vaginal Insert (MVI) 100 | Misoprostol Vaginal Insert (MVI) 50 | Cervidil 10 mg Vaginal Insert
Serious Adverse Events (participants affected / at risk) | 106/428 | 134/443 | 117/436
Other Adverse Events (participants affected / at risk) | 130/428 | 129/443 | 132/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol Vaginal Insert (MVI) 100 (N=428) | Misoprostol Vaginal Insert (MVI) 50 (N=443) | Cervidil 10 mg Vaginal Insert (N=436)
Arrested Labor (Pregnancy, puerperium and perinatal conditions) | 25 (25) | 36 (36) | 33 (33) — Also included terms such as Failure to progress
Cephalopelvic Disproportion (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 35 (35) | 29 (29)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abnormal Labor Affecting Fetus (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4) | 0 (0)
Foetal heart rate disorder (Pregnancy, puerperium and perinatal conditions) | 46 (46) | 47 (47) | 35 (35)
Foetal malpresentation (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 3 (3) | 6 (6)
Pregnancy-induced hypertension (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 5 (5)
uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1)
Liver abscess (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 2 (2) | 2 (2) | 3 (3)
cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
postpartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4) | 4 (4)
preeclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
uterine atony (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
bradycardia neonatal (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
tachcardia foetal (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
congenital anomaly (Congenital, familial and genetic disorders) | 10 (10) | 7 (7) | 7 (7)
Neonatal hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
hyperbilirubinemia neonatal (Hepatobiliary disorders) | 6 (6) | 5 (5) | 8 (8)
Group B sepsis neonatal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Apgar score low (Investigations) | 4 (4) | 2 (2) | 2 (2)
ABO hemolytic disease of the newborn (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 8 (9) | 3 (3)
cephalohaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
jaundice (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 1 (1)
neonatal aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
neonatal respiratory depression (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 5 (5)
neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 4 (4)
transient tachypnea of the newborn (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 4 (4)
infection prophylaxis (Surgical and medical procedures) | 2 (2) | 3 (3) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Misoprostol Vaginal Insert (MVI) 100 (N=428) | Misoprostol Vaginal Insert (MVI) 50 (N=443) | Cervidil 10 mg Vaginal Insert (N=436)
Abnormal labour affecting foetus (Pregnancy, puerperium and perinatal conditions) | 24 (24) | 12 (12) | 28 (28)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 30 (30) | 22 (22)
Foetal heart rate disorder (Pregnancy, puerperium and perinatal conditions) | 130 (130) | 129 (129) | 132 (132)
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 38 (38) | 45 (45) | 44 (44)
uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 83 (86) | 61 (63) | 81 (89)
uterine hypertonus (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 16 (16) | 25 (25)
Hypotension (Vascular disorders) | 18 (18) | 21 (21) | 23 (23)
Anemia (Blood and lymphatic system disorders) | 21 (21) | 25 (25) | 20 (20)
Perineal laceration (Pregnancy, puerperium and perinatal conditions) | 21 (21) | 28 (28) | 21 (21)
post partum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 16 (16) | 21 (21)
neonatal hyperbilirubinemia (Hepatobiliary disorders) | 9 (9) | 6 (6) | 15 (15)
Apgar score low (Investigations) | 10 (10) | 10 (10) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No